CLINICAL TRIAL: NCT06061575
Title: Comparison of the Efficacy of Paracetamol and Ibuprofen in the Management of Fever in Sepsis Patients: A Randomized Double-Blind Controlled Study
Brief Title: Comparison of the Efficacy of Paracetamol and Ibuprofen in the Management of Fever in Sepsis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Safa Dönmez, M.D., Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Management of Fever in Sepsis
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Sepsis; Acetaminophen; Fever; Ibuprofen
MeSH Terms: conditions — Sepsis; Fever | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetaminophen (Other): Adult patients diagnosed with sepsis according to the latest current guidelines, who have agreed to participate in the study or have provided consent by their relatives, and received 1g of acetaminophen for fever management.
  Interventions: Drug: Acetaminophen
- Ibuprofen (Other): Adult patients diagnosed with sepsis according to the latest current guidelines, who have agreed to participate in the study or have provided consent by their relatives, and received 400 mg of ıbuprofen for fever management.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Acetaminophen — fever will be managed with acetaminophen
  Other Names: Acetaminophen 1gr
  Arms: Acetaminophen
Drug: Ibuprofen — fever will be managed with ibuprofen
  Other Names: Ibuprofen 400 mg
  Arms: Ibuprofen

SUMMARY:
This is a randomized double-blind controlled study with the primary aim of scientifically evaluating the potential effects of paracetamol and ibuprofen in the management of sepsis by comparing their fever-reducing efficacy in septic patients. Sepsis is recognized as a severe form of systemic inflammatory response syndrome (SIRS) characterized by organ dysfunction resulting from severe infections. This study aims to address a significant aspect of fever management in septic patients by objectively assessing the fever-reducing potential of paracetamol and ibuprofen.

DETAILED DESCRIPTION:
This is a randomized double-blind controlled study with the primary aim of scientifically evaluating the potential effects of paracetamol and ibuprofen in the management of sepsis by comparing their fever-reducing efficacy in septic patients. Sepsis is recognized as a severe form of systemic inflammatory response syndrome (SIRS) characterized by organ dysfunction resulting from severe infections. This study aims to address a significant aspect of fever management in septic patients by objectively assessing the fever-reducing potential of paracetamol and ibuprofen.

In addition to assessing the fever-reducing efficacy of paracetamol and ibuprofen, this study will also evaluate their ability to provide symptomatic relief. The effects of paracetamol and ibuprofen on vital signs in septic patients will be examined to understand the overall course of the clinical condition. The analysis of the side effect profile aims to provide a comprehensive view of the safety and tolerability of both drugs.

The significance of this study can be explained by the critical role of fever regulation in sepsis management. Commonly used drugs like paracetamol and ibuprofen are widely employed to reduce fever and alleviate symptoms. However, there is limited data regarding the efficacy and safety of these drugs in septic patients. This research will help us better understand the role of these drugs in fever management in septic patients and contribute to optimizing treatment strategies. The findings of this study may guide clinical practice and establish a stronger scientific foundation for the management of septic patients.

This research may bring a new perspective to clinical practices regarding fever management in septic patients. By providing scientific data on whether commonly used drugs like paracetamol and ibuprofen can contribute to sepsis treatment, it may enhance the more effective management of patients. If it is demonstrated that paracetamol and ibuprofen can be used effectively and safely in septic patients, treatment optimization can be achieved with appropriate dosages and under suitable conditions. This may enable patients to achieve more effective fever control.

The results of the research may offer a better scientific basis for the use of drugs like paracetamol and ibuprofen in septic patients in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Under 80 years of age
* Willing to participate in the study
* Diagnosed with sepsis according to the latest current guidelines
* Having a fever >38.3°C
* With no known history of adverse reactions to the active ingredient of the medication to be used"

Exclusion Criteria:

* Under 18 years of age or over 80 years of age
* Not willing to participate in the study
* With a known history of adverse reactions to study medications
* Having a fever <38.3°C
* Pregnant individuals
* Individuals with advanced systemic illness
* Those with malignancies
* Patients with chronic liver and kidney disease
* Using sedative and analgesic neuro-psychiatric drugs
* With a history of psychological and neurological diseases"

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Fever | 30.-60.-120. minutes
  Body temperature, celcius

SECONDARY OUTCOMES:
Heart Rate | 30.-60.-120. minutes
  Heart rate per minute
Blood Pressure | 30.-60.-120. minutes
  Systolic and diastolic blood pressure in mmHg
Oxygen saturation | 30.-60.-120. minutes
  Measured as a percentage through capillary measurement

CONTACTS AND LOCATIONS:
Overall Officials: SAFA DÖNMEZ, M.D., Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After publication in a journal, the research will be shared with interested researchers and the editorial team of the published journal.
Supporting Information: Study Protocol, SAP
Time Frame: The data can be obtained from the researchers upon request after the research has been published.
Access Criteria: The editorial team of the journal and other researchers granted permission by the investigators.

REFERENCES:
- [Background] Selladurai S, Eastwood GM, Bailey M, Bellomo R. Paracetamol therapy for septic critically ill patients: a retrospective observational study. Crit Care Resusc. 2011 Sep;13(3):181-6. PMID 21880006
- [Background] Lee BH, Inui D, Suh GY, Kim JY, Kwon JY, Park J, Tada K, Tanaka K, Ietsugu K, Uehara K, Dote K, Tajimi K, Morita K, Matsuo K, Hoshino K, Hosokawa K, Lee KH, Lee KM, Takatori M, Nishimura M, Sanui M, Ito M, Egi M, Honda N, Okayama N, Shime N, Tsuruta R, Nogami S, Yoon SH, Fujitani S, Koh SO, Takeda S, Saito S, Hong SJ, Yamamoto T, Yokoyama T, Yamaguchi T, Nishiyama T, Igarashi T, Kakihana Y, Koh Y; Fever and Antipyretic in Critically ill patients Evaluation (FACE) Study Group. Association of body temperature and antipyretic treatments with mortality of critically ill patients with and without sepsis: multi-centered prospective observational study. Crit Care. 2012 Feb 28;16(1):R33. doi: 10.1186/cc11211. PMID 22373120
- [Background] Ye S, Xu D, Zhang C, Li M, Zhang Y. Effect of Antipyretic Therapy on Mortality in Critically Ill Patients with Sepsis Receiving Mechanical Ventilation Treatment. Can Respir J. 2017;2017:3087505. doi: 10.1155/2017/3087505. Epub 2017 Mar 12. PMID 28386165
- [Background] Drewry AM, Ablordeppey EA, Murray ET, Stoll CRT, Izadi SR, Dalton CM, Hardi AC, Fowler SA, Fuller BM, Colditz GA. Antipyretic Therapy in Critically Ill Septic Patients: A Systematic Review and Meta-Analysis. Crit Care Med. 2017 May;45(5):806-813. doi: 10.1097/CCM.0000000000002285. PMID 28221185
- [Background] Bernard GR, Wheeler AP, Russell JA, Schein R, Summer WR, Steinberg KP, Fulkerson WJ, Wright PE, Christman BW, Dupont WD, Higgins SB, Swindell BB. The effects of ibuprofen on the physiology and survival of patients with sepsis. The Ibuprofen in Sepsis Study Group. N Engl J Med. 1997 Mar 27;336(13):912-8. doi: 10.1056/NEJM199703273361303. PMID 9070471
- [Background] Haupt MT, Jastremski MS, Clemmer TP, Metz CA, Goris GB. Effect of ibuprofen in patients with severe sepsis: a randomized, double-blind, multicenter study. The Ibuprofen Study Group. Crit Care Med. 1991 Nov;19(11):1339-47. doi: 10.1097/00003246-199111000-00006. PMID 1935150
- [Background] Alaje EO, Udoh EE, Akande PA, Odey FA, Meremikwu MM. Ibuprofen versus paracetamol for treating fever in preschool children in Nigeria: a randomized clinical trial of effectiveness and safety. Pan Afr Med J. 2020 Aug 26;36:350. doi: 10.11604/pamj.2020.36.350.21393. eCollection 2020. PMID 33224416